CLINICAL TRIAL: NCT03281603
Title: A Study Comparing Patient Satisfaction and Retention of CAD /CAM Milled Complete Dentures and 3D Printed CAD/CAM Complete Dentures Versus Conventional Complete Dentures: A Randomized Clinical Trial
Brief Title: Patient Satisfaction & Retention of Milled, 3D Printed and Conventional Complete Dentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Abo Heikal, Assistant lecturer, Department of Prosthodontics, Faculty of Dentistry, MSA University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-08-24
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Complete Denture
Keywords: Patient satisfaction; Retention
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Masking Description: The Principal investigator, main supervisors and co-supervisor cannot be blinded as the trial will include digital designing of complete dentures on the CAD software and in the steps of the manufacturing techniques.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD/CAM complete denture (Experimental): First intervention: Constructing complete denture by CAD/CAM technology utilizing milling technique.
  Second intervention:Constructing complete denture CAD/CAM technology utilizing 3D printing technique
  Interventions: Device: CAD/CAM complete denture
- Conventional complete denture (Active Comparator): Constructing complete denture by conventional technique of denture processing
  Interventions: Device: CAD/CAM complete denture

INTERVENTIONS:
Device: CAD/CAM complete denture — complete denture will be designed by computer aided designing (CAD) and manufactured by computer aided manufacturing(CAM) utilizing Milling and 3D printing techniques

SUMMARY:
The objective of this trial is to compare patient satisfaction and retention of complete denture manufactured by three different techniques: CAD/CAM milling, CAD/CAM 3D printing and conventional technique.

DETAILED DESCRIPTION:
Patient examination and diagnosis will be made at the outpatient clinic, department of prosthodontics, faculty of Dentistry-Cairo University. Eligible Patients following the inclusion criteria will be consented to enrol in the trial. Randomization and allocation concealment will be done through sealed envelopes having groups for interventions and comparator. Each patient enrolled in the trial will pick an envelope having either the intervention or control group.

Preliminary impressions will be made and poured to study casts. Customizing trays from autopolymerising acrylic resins for final impressions with Zinc Oxide Eugenol , then impressions will be poured into dental stone producing master casts. Record bite blocks will then be constructed and bite registration will be made.

All bite records with their corresponding master casts will be digitalized by an extraoral desktop 3D scanner having the station sequence of scanning upper cast, lower cast then bite registration to be stored as standard triangulation language (STL) files.

STL files are then imported to EXOCAD design software designing full dentures with their permanent bases, teeth sizes and shapes following the recorded inter-arch space. Full upper and lower designed denture bases will be stored as STL files ready for manufacturing.

In first Intervention: STL files will be imported to SHERA CNC CAM software ready for nesting each file for the suitable PMMA block size and height, ready for milling them in denture bases with SHERA 5-axis Eco-mill milling machine . After milling denture bases, acrylic teeth will be chosen for each patient with the suitable shade and size following the inter-arch space, then glued by auto-polymerizing resin in their corresponding sockets in the milled denture bases.

In second intervention: STL files will be imported to Mogassam 3D-printer CAM software followed by adjusting the object to be virtually placed on X,Y and Z axes on the printer plate to be ready for layering it in three dimension. Photopolymerizable PMMA liquid resin will be added in the printer and the files processed into 3D printed upper and lower denture bases. Acrylic teeth are then glued in their sockets in the printed denture bases using auto-polymerizable resin.

In control group:Conventional complete denture construction by normal processing steps will be made for patients enrolled in the control group.

For the three groups, full dentures will be delivered and checked for occlusion, speech and mastication. Patient satisfaction will be assessed by a questionnaire template for each patient to be recorded at the day of delivery (baseline), 3months then 6 months. Retention for dentures will be assessed by engaging the snap hook on denture bases and pulling action will be made with the digital force gauge device to obtain the records on the day of delivery (baseline), 3months then 6 months' follow-up interval.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients ranging from age 55 to 75 years.
* Angle's Class I skeletal relationship.
* Well-developed ridge with U-shaped palatal vault and adequate firm mucosa.
* Last extraction took place six months ago.
* Normal facial symmetry.
* Cooperative patients.

Exclusion Criteria:

* -Temporomandibular disorders
* Uncontrolled diabetes
* Bleeding disorders or anticoagulant therapy
* Flabby tissues or sharp mandibular residual ridge.
* Heavy smokers.
* Patient's with neuromuscular disorders
* Patients on chemotherapy or radiotherapy
* Severe psychiatric disorders
* Angle's class II and III skeletal relationship

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | 6 months
  The questionnaire will include 5 main categories; each category having questions about Functional complaint about the denture, Overall mastication ability, Masticating ability for different types of food, Effect of mental and daily life and Overall denture satisfaction.

SECONDARY OUTCOMES:
Retention | 6 months
  Digital Force gauge device applying a pulling action on a snap hook attached to geometric center of denture bases

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M. Abo Heikal, PHD, Principal Investigator — Assistant lecturer, faculty of Dentistry, MSA University
Locations (2):
- Egypt (2):
  - Faculty of Dentistry,Cairo university, Giza
  - Cairo university, Giza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bidra AS, Taylor TD, Agar JR. Computer-aided technology for fabricating complete dentures: systematic review of historical background, current status, and future perspectives. J Prosthet Dent. 2013 Jun;109(6):361-6. doi: 10.1016/S0022-3913(13)60318-2. PMID 23763779
- [Background] Kanazawa M, Inokoshi M, Minakuchi S, Ohbayashi N. Trial of a CAD/CAM system for fabricating complete dentures. Dent Mater J. 2011;30(1):93-6. doi: 10.4012/dmj.2010-112. Epub 2011 Jan 26. PMID 21282882
- [Background] Maeda Y, Minoura M, Tsutsumi S, Okada M, Nokubi T. A CAD/CAM system for removable denture. Part I: Fabrication of complete dentures. Int J Prosthodont. 1994 Jan-Feb;7(1):17-21. PMID 8179777
- [Background] Han W, Li Y, Zhang Y, Lv Y, Zhang Y, Hu P, Liu H, Ma Z, Shen Y. Design and fabrication of complete dentures using CAD/CAM technology. Medicine (Baltimore). 2017 Jan;96(1):e5435. doi: 10.1097/MD.0000000000005435. PMID 28072686
- [Background] Infante L, Yilmaz B, McGlumphy E, Finger I. Fabricating complete dentures with CAD/CAM technology. J Prosthet Dent. 2014 May;111(5):351-5. doi: 10.1016/j.prosdent.2013.10.014. Epub 2014 Jan 23. PMID 24461946
- [Background] Chen H, Wang H, Lv P, Wang Y, Sun Y. Quantitative Evaluation of Tissue Surface Adaption of CAD-Designed and 3D Printed Wax Pattern of Maxillary Complete Denture. Biomed Res Int. 2015;2015:453968. doi: 10.1155/2015/453968. Epub 2015 Oct 25. PMID 26583108
- [Background] Inokoshi M, Kanazawa M, Minakuchi S. Evaluation of a complete denture trial method applying rapid prototyping. Dent Mater J. 2012 Feb 3;31(1):40-6. doi: 10.4012/dmj.2011-113. Epub 2012 Jan 21. PMID 22277604
- [Background] Torabi K, Farjood E, Hamedani S. Rapid Prototyping Technologies and their Applications in Prosthodontics, a Review of Literature. J Dent (Shiraz). 2015 Mar;16(1):1-9. PMID 25759851
- [Background] AlHelal A, AlRumaih HS, Kattadiyil MT, Baba NZ, Goodacre CJ. Comparison of retention between maxillary milled and conventional denture bases: A clinical study. J Prosthet Dent. 2017 Feb;117(2):233-238. doi: 10.1016/j.prosdent.2016.08.007. Epub 2016 Oct 17. PMID 27765399
- [Background] Bilhan H, Erdogan O, Ergin S, Celik M, Ates G, Geckili O. Complication rates and patient satisfaction with removable dentures. J Adv Prosthodont. 2012 May;4(2):109-15. doi: 10.4047/jap.2012.4.2.109. Epub 2012 May 30. PMID 22737317